CLINICAL TRIAL: NCT05430672
Title: A Prospective, Multicenter, Objective Performance Criteria-Controlled Study for National Medical Products Administration Approval Of The Thoracic Aortic Stent Graft System
Brief Title: Safety and Efficacy Study Of The Thoracic Aortic Stent Graft System Treating Aortic Dissection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zhejiang Zylox Medical Device Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: V1.1/2021-11-16
Record Dates: First submitted 2022-01-25; First posted 2022-06-24 (Actual); Last update posted 2022-06-24 (Actual); Status verified 2022-01

CONDITIONS: Aortic Dissection
Keywords: Aortic Dissection; Thoracic aortic; Stent graft
MeSH Terms: conditions — Aortic Dissection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Subjects with aortic dissection (Other): Subjects receive endovascular treatment.
  Interventions: Device: The Thoracic Aortic Stent Graft System (Zylox-Tonbridge Medical Technology Co., Ltd. )

INTERVENTIONS:
Device: The Thoracic Aortic Stent Graft System (Zylox-Tonbridge Medical Technology Co., Ltd. ) — This is a objective performance criteria-controlled study, all subjects meet the criteria will receive the same treatment using the thoracic aortic stent graft system (Zylox-Tonbridge Medical Technology Co., Ltd. ).

SUMMARY:
This is a prospective, multicenter and single-arm trail to study the safety and efficacy of the thoracic aortic stent graft system that specially designed for treating aortic dissection.

DETAILED DESCRIPTION:
This trail is conducted in several centers all around China. In about 18 months, 120 subjects with aortic dissection will be recruited, all of which receive endovascular treatment using the thoracic aortic stent graft system (Zylox-Tonbridge Medical Technology Co., Ltd. ). The subjects will be followed up in 30 days/ 6 months/ 12 months/ 2-5 years.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 80 years;
* Subject or legal representative is able to understand the purpose of study, agrees to comply with protocol requirements and has provided written informed consent；
* Subjects who are diagnosed with Stanford type B aortic dissection requiring reconstruction of the left common carotid artery and left subclavian artery or requiring reconstruction of the left subclavian artery;
* Appropriate access to the femoral artery, iliac artery, brachial artery, etc. that can be used for endoluminal aortic therapy.

Exclusion Criteria:

* The same surgery requires intervention for other vascular lesions；
* History of surgery in the aortic arch or endovascular repair surgery;
* Severe stenosis or calcification or distortion in the anchoring area of the proximal end of the stent;
* Subjects with severe liver, kidney failure；
* Subjects with severe coagulation disorders；
* Female subjects who are pregnant, lactating within the study period or unable to contraception during the trail.
* History of allergies to anesthetics, contrast agents or the material of stent/ deliver system；
* Inability to tolerate anesthesia；
* History of acute myocardial infarction, cerebral infarction or cerebral hemorrhage within 3 months before surgery;
* Subjects who have participated in any other drug or medical device clinical investigations and haven't reach the primary endpoint.
* Subjects with acute systemic infection
* Other circumstances judged by researchers that are not suitable for enrollment .

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-06 (Estimated); Primary Completion 2023-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Rate of no Major Adverse Event (MAE) | Immediately after the intervention
  MAE was defined as aortic dissection related death, disabling stoke or paraplegic.
Rate of no Major Adverse Event (MAE) | 30 days
  MAE was defined as aortic dissection related death, disabling stoke or paraplegic.
Success rate of endovascular treatment | Up to 12 months
  * Technique success: the delivery system was successfully delivered to the predetermined position, the stent was accurately positioned and successfully deployed, and the delivery system could be safely withdrawn from the body, no type I or type III endoleak can be found during angiography.
  * No stent displacement during 12 months follow up time.
  * No secondary surgical intervention during 12 months follow up.

SECONDARY OUTCOMES:
Rate of aortic dissection related mortality | Intraoperation/ 30 days/ 6 months/ 12 months/ up to 2-5 years
  Death caused by aortic dissection rupture or related treatment.
Rate of all cause mortality | Intraoperation/ 30 days/ 6 months/ 12 months/ up to 2-5 years
  Death for any reason will be recorded.
Rate of Adverse Events(AE) | Intraoperation/ 30 days/ 6 months/ 12 months/ up to 2-5 years
  The definition of AE(Adverse Event) refers to International Organization for Standardization (ISO) 14155, AE should be distinguished from normal postoperative stress response.
Rate of Serious Adverse Events(SAE) | Intraoperation/ 30 days/ 6 months/ 12 months/ up to 2-5 years
  The definition of SAE (Serious Adverse Event) refers to ISO 14155.
Rate of technique success | Immediately after the intervention
  The delivery system was successfully delivered to the predetermined position, the stent was accurately positioned and successfully deployed, and the delivery system could be safely withdrawn from the body, no type I or type III endoleak can be found during angiography.
Incidence of stent displacement | 30 days/ 6 months/ 12 months
  Stent displacement was defined as the aortic and branch stent-grafts displacing by more than 10 mm from the post-implantation position.
Success rate of endovascular repair | 30 days/ 6 months/ 12 months
  Comparison of CTA results before surgery and within 30 days, 6 months, and 12 months after surgery. Changes in the diameter of the stent covered by aortic dissection and thrombosis of the false lumen are used to determine whether the vessel is successfully repaired.

CONTACTS AND LOCATIONS:
Overall Officials: Xinwu Lu, Principal Investigator — Shanghai Ninth People's Hostpital, Shanghai JiaoTong University School of Medicine
Locations (14):
- China (14):
  - The First Affiliated Hospital of Bengbu medical College, Bengbu, Anhui
  - The Second Hospital Of Anhui Medical University, Hefei, Anhui
  - Liuzhou Worker's Hospital, Liuchow, Guangxi
  - Huaihe Hospital of Henan University, Kaifeng, Henan
  - The First Affiliated Hospital Of Zhengzhou University, Zhengzhou, Henan
  - Renmin Hospital Of Wuhan University, Wuhan, Hubei
  - Nanjing Drum Tower Hospital, the affiliated Hospital of Nanjing University Medical School, Nanjing, Jiangsu
  - The Second Affiliated Hospital Of Nanchang University, Nanchang, Jiangxi
  - The First Affiliated Hospital of Xi'An Jiaotong University, Xi'an, Shaanxi
  - The First Hospital Of Zhejiang Province, Hanzhou, Zhejiang
  - The First Affiliated Hospital Of WMU, Wenzhou, Zhejiang
  - Peking Union Medical College Hospital, Beijing
  - Shanghai Ninth People's Hostpital, Shanghai JiaoTong University School of Medicine, Shanghai
  - Zhongshan Hospital, Shanghai